CLINICAL TRIAL: NCT00647998
Title: Phase 2 Dose Finding Trial of Prophylactic Darbepoetin Alfa to Improve Outcomes From Ischemic Complications of Surgery
Brief Title: The Darbepoetin Alfa for Ischemic Surgical Complications (DISC) Dose Finding Trial
Acronym: DISC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Steven Messe, Associate professor of neurology, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DISC-001
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Spinal Ischemia; Stroke; Neuroprotection
Keywords: Surgical complications; Spinal ischemia; Stroke; Neuroprotection
MeSH Terms: conditions — Stroke | interventions — Darbepoetin alfa; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Darbepoetin (Experimental): Patients received 1mg/kg IV Darbepoetin immediately prior to surgery
  Interventions: Drug: Darbepoetin alfa; Other: Standard care
- Standard care (Placebo Comparator): No Darbepoetin
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: Darbepoetin alfa — Patients will receive one IV injection of Darbepoetin alfa at doses ranging from 1mcg/kg to 6.5 mcg/kg prior to surgery
  Other Names: Aranesp
  Arms: Darbepoetin
Other: Standard care

SUMMARY:
Numerous neuroprotectants have been effective when given prior to ischemic stroke in animals, yet they have all have failed when given after ischemic stroke in humans. A novel approach to ischemic neuroprotection is needed. Many patients who undergo cardiac, vascular, and neurosurgical procedures develop ischemic central nervous system (CNS) complications. These high risk surgeries present a unique opportunity to administer neuroprotectant medication prior to the injury, greatly increasing the likelihood that it will have a positive impact on outcomes. Patients undergoing descending thoracic aortic (DTA) and thoracoabdominal aortic (TAA) surgery have a particularly high rate of both brain and spine ischemia. In addition, these surgeries require placement of a lumbar cerebrospinal fluid (CSF) drain, allowing access to CSF in order to monitor markers of injury and penetration of medication into the CNS. We are performing a pilot dose finding trial of prophylactic darbepoetin alfa, a long-acting erythropoiesis medication with putative neuroprotectant properties, in patients undergoing DTA and TAA surgery.

DETAILED DESCRIPTION:
Numerous neuroprotectants have been effective when given prior to ischemic stroke in animals, yet they have all have failed when given after ischemic stroke in humans. A novel approach to ischemic neuroprotection is needed. Many patients who undergo cardiac, vascular, and neurosurgical procedures develop ischemic central nervous system (CNS) complications. These high risk surgeries present a unique opportunity to administer neuroprotectant medication prior to the injury, greatly increasing the likelihood that it will have a positive impact on outcomes. Patients undergoing descending thoracic aortic (DTA) and thoracoabdominal aortic (TAA) surgery have a particularly high rate of both brain and spine ischemia. In addition, these surgeries require placement of a lumbar cerebrospinal fluid (CSF) drain, allowing access to CSF in order to monitor markers of injury and penetration of medication into the CNS. We performed a pilot dose finding trial of prophylactic darbepoetin alfa, a long-acting erythropoiesis medication with putative neuroprotectant properties, in patients undergoing DTA and TAA surgery. This dose finding trial was stopped early after 9 patients were enrolled at the request of the FDA after an unrelated trial of erythropoietin in acute stroke performed in Germany was negative and showed possible harm in those patients who received intravenous tissue plasminogen activaor (tPA). We then enrolled 9 additional patients who did not receive any intervention in order to compare them to the patients who received darbepoetin.

ELIGIBILITY:
Inclusion Criteria:

* Are men and women between the ages of 18 - 100 years old (inclusive)
* Require descending thoracic or thoracoabdominal aorta surgical repair
* Can provide informed consent

Exclusion Criteria:

* Have a traumatic aortic dissection
* Have a baseline NIHSS > 1 or modified Rankin Scale > 1
* Have a history of stroke or myocardial infarction within the past 30 days
* Have a preoperative hemoglobin < 9 or > 14
* Have a history of polycythemia vera or essential thrombocytosis
* Have a history of hematologic malignancy
* Have a history of arterial or venous thrombosis in the past three months
* Have uncontrolled hypertension
* Have active malignancy requiring treatment
* Are receiving hemodialysis
* Are currently using recombinant human erythropoietin or darbepoetin alfa, or have an expectation to require these medications within 30 days of surgery.
* Have a known allergy to recombinant human erythropoietin or darbepoetin alfa
* Are pregnant or breast-feeding. Women of childbearing potential must have a negative pregnancy test (urine pregnancy test or serum beta-HCG)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Messe SR, McGarvey ML, Bavaria JE, Pochettino A, Szeto WY, Cheung AT, Leitner E, Miller SW, Kasner SE. A pilot study of darbepoetin alfa for prophylactic neuroprotection in aortic surgery. Neurocrit Care. 2013 Feb;18(1):75-80. doi: 10.1007/s12028-012-9710-4. PMID 22528284

RESULTS

PARTICIPANT FLOW:
Groups:
- Darbepoetin Alfa: Patients receive 1 mg/kg IV darbepoetin immediately before surgery
Period: Overall Study
Arm/Group | Darbepoetin Alfa | Standard Care
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Darbepoetin Alfa | Standard Care | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [55 to 67] | 62 [58 to 64] | 59 [55 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
Prior stroke [Count of Participants; unit: Participants] | 3 | 3 | 6
Prior aortic surgery [Count of Participants; unit: Participants] | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Death or Neurologic Disability, Defined as an National Institutes of Health Stroke Scale (NIHSS)>4 or American Spinal Injury Association (ASIA) Lower Extermity Motor Score <25
Description: The NIHSS is a validated quasi-ordinal measure of stroke severity. An NIHSS >4 is generally considered moderate or severe. The ASIA Lower Extremity Motor Score is a cumulative total of assessments of strength in 5 muscles in each leg, using the Medical Research Council 0-5 stroke score. ASIA score < 25 is associated with impaired ambulation.
Time Frame: Discharge from the hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin Alfa | Standard Care
Number analyzed (Participants) | 9 | 9
Participants | 1 | 3

2. Secondary Outcome: CSF S100beta
Description: Cerebrospinal fluid S100beta level
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- Darbepoetin: Patients received 1mg/kg IV Darbepoetin immediately prior to surgery
  Darbepoetin alfa: Patients will receive one IV injection of Darbepoetin alfa at doses ranging from 1mcg/kg to 6.5 mcg/kg prior to surgery
  Standard care
- Standard Care: No Darbepoetin
  Standard care
Arm/Group | Darbepoetin | Standard Care
Number analyzed (Participants) | 9 | 9
pg/mL | 214 [118 to 235] | 260 [68 to 1175]

3. Secondary Outcome: Hemoglobin
Time Frame: 24 hours post-surgery
Measure: Mean (Standard Deviation); unit: gm/dL
Arm/Group | Darbepoetin Alfa | Standard Care
Number analyzed (Participants) | 9 | 9
gm/dL | 10.4 (2.1) | 9.5 (0.7)

ADVERSE EVENTS:
Arm/Group | Darbepoetin Alfa | Standard Care
Serious Adverse Events (participants affected / at risk) | 4/9 | 3/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa (N=9) | Standard Care (N=9)
Spinal ischemia (Nervous system disorders) | 2 | 1
Stroke (Nervous system disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No